CLINICAL TRIAL: NCT04489836
Title: GlutDigest - Enzymes-assisted Gluten Digestion (Pilot Study)
Brief Title: GlutDigest - Pilot Study
Acronym: GlutDigestP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deerland Enzymes (Industry)
Collaborators: Teagasc (Industry); Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Project 0470-Pilot study
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Main Focus: Gluten and Starch Digestibility
Keywords: Gluten; Starch; Digestive enzymes; Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal A + Glutalytic® (Experimental): 350 mg Glutalytic® capsule, taken by mouth, once, with Meal A
  Interventions: Dietary Supplement: Glutalytic®; Other: Meal A
- Meal A + DE111® (Experimental): 350 mg DE111® capsule, taken by mouth, once, with Meal A
  Interventions: Dietary Supplement: DE111®; Other: Meal A

INTERVENTIONS:
Dietary Supplement: Glutalytic® — Glutalytic® capsule
  Arms: Meal A + Glutalytic®
Dietary Supplement: DE111® — DE111® capsule
  Arms: Meal A + DE111®
Other: Meal A — Oatmeal porridge - serving of oat porridge (cooked) containing 50g of carbohydrates (excluding sugars); Wheat cereal - serving of wheat cereal providing 1g of gluten; Water - 125 mL

SUMMARY:
This is a pilot, feasibility study to evaluate, test and optimize sample analysis procedures and protocols before the full-scale, crossover study is conducted.

DETAILED DESCRIPTION:
Two important factors can influence the proportions of gluten and starch that resist digestion: (1) enzyme availability and specificity and (2) the structural properties of the food. A complete evaluation of gluten digestion and of the impact of dietary supplements is difficult to conduct because it is not easy to obtain samples of digestive chime. The analysis of the ileal effluent of healthy ileostomy patients constitutes a non-invasive alternative to intubation techniques for the study of nutrient digestion and of the fate of probiotics in the small intestine.

The main aim of this study is to test and optimize sample analysis protocols before conducting the full-scale, crossover study which will aim at evaluating the impact of two dietary supplements (Glutalytic® and DE111®) and of oatmeal properties on the digestion of gluten and starch and on the glycemic response.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent
* Subject has an ileostomy stable for at least 3 months post-operative and shows normal stoma functions
* Subject is otherwise healthy
* Subject is available to participate in the study sessions on the proposed dates

Exclusion Criteria:

* Subject has coeliac disease or allergy to wheat products and/or any other ingredients in the test meal and standard meals
* Case of obstruction of the stoma in the past 3 months
* Body mass index < 18 kg/m2 or > 30 kg/m2.
* Diagnosed mouth, throat or active gastrointestinal pathology (other than ileostomy) that may affect normal ingestion and digestion of food.
* History of pancreatic disease
* Subject is immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year)
* Subject has Type 1 or Type 2 diabetes mellitus.
* Subject has a history of bariatric surgery.
* Subject has a history of drug and/or alcohol abuse at the time of enrolment
* Subject is currently participating in another study, or plans to participate in another study during the study period
* Women of child-bearing potential who do not use an acceptable method of contraception
* Pregnant or nursing (lactating) women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-09-19 (Actual); Study Completion 2020-09-19 (Actual)

PRIMARY OUTCOMES:
Undigested wheat protein after each treatment | 9-hour period after the test meal
  Difference between the mean concentration of undigested wheat protein in ileal effluent samples.

SECONDARY OUTCOMES:
Vegetative DE111 cells | 9-hour period after the test meal
  Mean concentration of DE111® cells recovered in the ileal effluent samples.
Glycemic response | At baseline, and at different time-points in the 9-hour period after consumption of the test meal.
  Difference between the mean area under the glucose concentration (measured in the interstitial fluid) curves following each treatment.
Undigested starch | 9-hour period after the test meal
  Difference between the mean concentration of undigested starch in ileal effluent samples.
Undigested food particles | 9-hour period after the test meal
  Pictures of undigested foods particles and microscopy will be combined for a combined assessment of macro- and micro- structural characteristics of the food particles recovered in ileal effluent samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No